CLINICAL TRIAL: NCT03330834
Title: Safety and Toxicity of CAR-T Cell Immunotherapy in Patients With Advanced Lung Cancer After Standard Treatment Failure: A Single-Arm and Single-Center Phase I Clinical Study
Brief Title: CAR-T Cell Immunotherapy for Advanced Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Serious adverse events
Sponsor: Sun Yat-sen University (Other)
Collaborators: Guangzhou Yiyang Biological Technology Co., Ltd. (Other)
Responsible Party: Principal Investigator, Li Zhang, MD, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CART-YY2017
Record Dates: First submitted 2017-10-01; First posted 2017-11-06 (Actual); Results first posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Advanced Lung Cancer
Keywords: CAR-T; advanced lung cancer; single-arm; phase I clinical study

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): CAR-T cells to treat advanced lung cancer. This study has only one arm. All participators will attend the screening and meet the set criteria for the clinical treatment. PD-L1 CAR-T cells are infused on day 0 with 10%, day 3 with 30% and day 7 with 60% , (1-2)×10^6/kg PD-L1 CAR-T cells total.
  Interventions: Biological: CAR-T cells to treat advanced lung cancer

INTERVENTIONS:
Biological: CAR-T cells to treat advanced lung cancer — Drug: fludarabine. On days -4 through -2, fludarabine (25mg/m2) will be infused for 3 consecutive days; Drug: cyclophosphamide. On days -4 through -2, cyclophosphamide (250mg/m2) will be infused for 3 consecutive days.
  Patients will receive the above chemotherapy for lymphocyte-depletion followed by PD-L1 CAR-T cells.

SUMMARY:
The NSCLC patients who failed the standard treatments, with positive Programmed Death-Ligand 1 (PD-L1) expression, were enrolled into this trial. About 22 advanced NSCLC patients will be screened according to the criteria. The qualified patients will be recruited and sign the informed consent.Participants will be hospitalized and undergo clinical examinations.

Appropriate volume of peripheral blood will be draw (from 66 ml to 360 ml, depend on the body weight and blood routine test), using Ficoll method to centrifuge peripheral blood cell and collected T cells. PD-L1 CAR gene is cloned in a lenti-viral vector that was composed of T cell activation molecules (Cluster of Differentiation 137 (CD137/CD28) and Cluster of Differentiation 3(CD3) zeta intracellular domains) and PD-L1 single-chain variable fragment(scFv) derived from the variable regions of a PD-L1 monoclonal antibody.Then, investigators packaged pseudo-lentiviral particles in human embryonic kidney (293T) cells that will be used to transduce autologous T cells isolated from the patients. CAR positive T lymphocytes will be determined by FACS with florescence labeled goat anti-human F(ab')2. The plasmids, pseudo-lentiviral particles and transduced T cells will be subject to the stipulated tests by a third party.

Patients will receive leukodepletion chemotherapy (cyclophosphamide: 250mg/m^2 × 3 days; fludarabine: 25mg/m^2× 3 days). One day later, the chemotherapeutic effects would be assessed. PD-L1 CAR-T cells will be infused on day 0 with 10%, day 3 with 30% and day 7 with 60% (total number is (1-2)×10^6/kg). The patients will be observed closely for any adverse reactions and if happened, given supportive treatments.

The patients will be discharged on day 14 and will be followed up for two years according to the study scheme, i.e. once a month for the first three months; once every two months in the first year; since then, once a quarter in the second year. The persistence of PD-L1 CAR-T cells in the circulation will be monitored by fluorescent activated cell sorting (FACS) and polymerase chain reaction (PCR). If the patients undergo core needle biopsy, the infiltration of CAR positive cells in the tumor tissue will be evaluated by immunohistochemistry (IHC). The safety profile and anti-tumor efficacy of the CAR-T cells immunotherapy will be assessed during the whole process based on CTCAE v4.1 and RECIST v1.1.

DETAILED DESCRIPTION:
The morbidity and mortality of lung cancer ranks the first in all malignancies. Although targeted therapy such as epidermal growth factor receptor (EGFR) tyrosine kinase inhibitors (TKI) and activated lymphocyte kinase (ALK)-TKI can prolong non-small cell lung cancer (NSCLC) patients' survival, drug resistance almost occurs inevitably.

In recent years, PD-L1/PD-1 antibodies like Nivolumab and Pembrolizumab, show satisfactory therapeutic potential in the treatment of cancers like melanoma and lung cancer. Latest clinical investigations show that anti-PD-1 or PD-L1 antibody therapy can prolong patients' survival but actually only 20% of patients benefited from it.

Chimeric antigen receptor T-Cell (CAR-T) was genetically modified T lymphocytes by pseudo-lentiviral transduction to provide them with high binding affinity and specificity to the tumor antigen. That affinity was provided by CAR, independent from major histocompatibility complex (MHC).

CAR-T cell immunotherapy had shown tremendous success in the treatment of acute lymphocytic leukemia (ALL). Cluster of Differentiation (CD)-19 CAR-T cell treatment archived as high as 92% complete response rate for refractory and recurrent ALL. When the CAR-T cells targeting Her2/neu were given to the patients, mortality was observed from cardiopulmonary failure due to the weak expression of Her2/neu on the pulmonary epithelial cells. In contrast, Her2/neu antibody (trastuzumab) is widely applied safely in clinic to treat breast cancer patients. It strongly suggests that the CAR-T cells are more potent.

Thus investigators hypothesized that the CAR targeting tumor cell PD-L1 would significantly improve the efficacy of CAR-T cells and extend their application in the treatment of solid tumors, especially lung cancer. Investigators designed and cloned a PD-L1 CAR gene that targets the PD-L1 expressed on tumor cells. Given that PD-L1 CAR-T cells can effectively kill not only PD-L1 positive tumor cells in vivo but also immunosuppressive cells (like myeloid-derived suppressor cells (MDSCs)) inside tumors, they can remarkably improve immunosuppressive tumor microenvironment. Accordingly they can restore the function of tumor infiltrated T-lymphocytes(TILs) to achieve the synergistic effect of killing tumor cells that can greatly enhance the killing effects of PD-L1 CAR-T cells on tumor cells, even eliminate tumors.

The preclinical studies showed that PD-L1 CAR-T cells could be activated by and had significant killing effects on PD-L1 positive tumor cells in vitro. They inhibited tumor growth, while no obvious toxicity have been observed in mouse xenograft models. Investigators decide to explore the safety and efficacy of the new CAR-T cells in the phase I clinical study in the treatment of advanced NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects were diagnosed with NSCLC by pathology and at clinical stages ⅢB/Ⅳ based on the 8th Union for International Cancer Control/American Joint Committee on Cancer (UICC/AJCC) Staging System or the disease has recurred or progressed after multi-mode therapy (radiotherapy, surgical excision or radical radiotherapy/chemotherapy to treat local advanced lesions ).
2. Subjects whose recurrent or advanced NSCLC has progressed after standard treatments (operation, radiotherapy and targeting therapy, not including PD-1/PD-L1 checkpoint inhibition therapy) or who are reluctant to receive chemotherapy.
3. Subjects should undertake core needle biopsy again to collect at least one fresh biopsy specimen and at least 10 non-stained sections before recruitment.
4. TKI or chemotherapeutic should be discontinued at least 21 days before Day 0 of the clinical trial while radiotherapy of lung cancer at least 6 months before Day 0 of the clinical trial . Subjects should receive baseline imaging scan after the previous treatments are suspended.
5. Lesions must be detected by CT or MRI according to RECIST 1.1 Criteria. Tumor imaging should be performed at least within 28 days before the beginning of the clinical study.
6. Age>=18 years old and weight >=40kg.
7. PD-L1 is positive by IHC in tissue biopsies of progressive lung cancer after standard treatments(>10%).Ventana PD-L1 (SP142) approved by FDA is used to detect PD-L1 expression level on participated patients' lung cancer sections.
8. Life expectancy>=12 weeks
9. Eastern Cooperative Oncology Group (ECOG) score≤ 2
10. Blood pregnancy tests should be negative within 14 days before the woman of childbearing age starts treatment and agrees to take contraceptive methods with a failure rate of no more than 1% per year until the final follow-up.Contraceptive methods with a failure rate of no more than 1% per year include tubal ligation, vasectomy, hormonal contraceptives, intrauterine hormone release system and copper intrauterine device (IUDs).
11. Hematology and liver and kidney functions should meet the following laboratory values. These laboratory tests should be completed in 7 days before the first therapeutic cell infusion.

    Tests and Laboratory Values:

    Hematology:
    1. White Blood Cell (WBC): >=3.5*10^9/L;
    2. Absolute Neutrophil Count (ANC): >=1.5*10^9/L;
    3. Hemoglobin (HGB): >=90g/L;
    4. Platelet (PLT): >=80*10^9/L;

    Blood Coagulation Function:

    PT、APTT、FIB、TT: within normal limits;

    Liver Function:
    1. Aspartic Transaminase (AST): <2.5*upper normal limits(ULN)(hepatic metastasis subjects with 0-1 ECOG score < 5*ULN);
    2. Alanine Aminotransferase (ALT): <2.5*ULN(hepatic metastasis subjects with 0-1 ECOG scorer < 5*ULN);
    3. Total Bilirubin (TIBC): <1.5*ULN;

    Kidney Function:

    Serum Creatinine (CR): <1.0*ULN.
12. Subjects are willing to participate in this study and agree to sign the Informed Consent.

Exclusion Criteria:

1. Subjects who are receiving systematic steroid treatments 3 days before the first cell treatment.

   Notice:
   1. Corticosteroids can be used to treat adverse event (AE) and serious adverse event (SAE) after the experimental cell treatment.
   2. Subjects who receive steroid replacement therapy everyday can be included in the clinical study. Prednisone therapy in a dose of 5-7.5mg/day is replacement therapy.
   3. Subjects who receive equivalent dose of hydrocortisone treatment as replacement therapy are also allowed into the clinical trial.
2. Subjects who have received systematic cytotoxic chemotherapy, biological therapy or major operations in 3 weeks before the first dose of experimental cell therapy or subjects who have received lung radiation more than 30 gray (Gy) in 6 months before the first dose of experimental cell therapy.
3. Subjects who have received previous cell treatments such as CAR-T and cytokine-induced killer (CIK) cells or anti-PD-1 or anti- PD-L1 antibody treatment.
4. Subjects with confirmed Central Nervous System (CNS) metastasis and/or carcinomatous meningitis.

   Notice:

   Subjects who have received brain metastasis treatments are allowed in this study, in the case that subjects' conditions are stable (no CNS symptoms) and no radiographic evidence of new or extensive brain metastasis is found at least 4 weeks after the treatments (such as operation or RT). Subjects should suspend hormone treatment at least 3 days before the first dose of experimental cell treatment.
5. Subjects with active autoimmune diseases who need systematic treatments (such as disease improving drugs, corticosteroids and immunosuppressive drugs) in the last 2 years.

   Notice:

   Replacement therapy (thyroxine, insulin or physiological corticosteroid replacement therapy to treat adrenal dysfunction or pituitary dysfunction) is not considered as systematic therapy. Subjects who need inhalation corticosteroid therapy can be included in this trial. Subjects with vitiligo or in long-term remission of pediatric asthma or allergic diseases can be included in this trial.
6. Subjects with interstitial pneumonia or a history of pneumonia with oral or intravenous steroid treatments.
7. Subjects whose lymphocytes are difficult to transduce (<20%) or can not proliferate over 5 times.
8. Subjects who have received allotransplantation or solid organ transplantation.
9. Subjects who have received or will receive live vaccines in 30 days before the first experimental cell treatment. Inactivated seasonal flu vaccination is allowed.
10. Subjects with active infections who need intravenous systematic treatments.
11. Subjects with a history of human immunodeficiency virus (HIV)（HIV 1/2 antibody positive）infection.
12. Subjects with known active hepatitis B or hepatitis C. Subjects with HBsAg positive will be excluded. The definition of active hepatitis C is that hepatitis C antibody is positive while quantitative hepatitis C virus (HCV) RNA results exceed the lower detection limit.
13. Subjects with a history of mental disorders or drug abuse that may influence treatment compliance.
14. Women in pregnancy or lactation or are expected to be pregnant during the study (from the screening and to 60 days after the final experimental cell treatment) or men whose wives are in pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2020-04-14 (Actual); Study Completion 2020-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Landis SH, Murray T, Bolden S, Wingo PA. Cancer statistics, 1999. CA Cancer J Clin. 1999 Jan-Feb;49(1):8-31, 1. doi: 10.3322/canjclin.49.1.8. PMID 10200775
- [Background] Novello S, Le Chevalier T. Chemotherapy for non-small-cell lung cancer. Part 1: Early-stage disease. Oncology (Williston Park). 2003 Mar;17(3):357-64. PMID 12661267
- [Background] Ettinger DS, Wood DE, Akerley W, Bazhenova LA, Borghaei H, Camidge DR, Cheney RT, Chirieac LR, D'Amico TA, Demmy TL, Dilling TJ, Govindan R, Grannis FW Jr, Horn L, Jahan TM, Komaki R, Kris MG, Krug LM, Lackner RP, Lanuti M, Lilenbaum R, Lin J, Loo BW Jr, Martins R, Otterson GA, Patel JD, Pisters KM, Reckamp K, Riely GJ, Rohren E, Schild S, Shapiro TA, Swanson SJ, Tauer K, Yang SC, Gregory K, Hughes M. Non-small cell lung cancer, version 1.2015. J Natl Compr Canc Netw. 2014 Dec;12(12):1738-61. doi: 10.6004/jnccn.2014.0176. PMID 25505215
- [Background] Sholl LM, Aisner DL, Varella-Garcia M, Berry LD, Dias-Santagata D, Wistuba II, Chen H, Fujimoto J, Kugler K, Franklin WA, Iafrate AJ, Ladanyi M, Kris MG, Johnson BE, Bunn PA, Minna JD, Kwiatkowski DJ; LCMC Investigators. Multi-institutional Oncogenic Driver Mutation Analysis in Lung Adenocarcinoma: The Lung Cancer Mutation Consortium Experience. J Thorac Oncol. 2015 May;10(5):768-777. doi: 10.1097/JTO.0000000000000516. PMID 25738220
- [Background] Pardoll DM. The blockade of immune checkpoints in cancer immunotherapy. Nat Rev Cancer. 2012 Mar 22;12(4):252-64. doi: 10.1038/nrc3239. PMID 22437870
- [Background] Johnson DB, Sosman JA. Therapeutic Advances and Treatment Options in Metastatic Melanoma. JAMA Oncol. 2015 Jun;1(3):380-6. doi: 10.1001/jamaoncol.2015.0565. PMID 26181188
- [Background] Garon EB, Rizvi NA, Hui R, Leighl N, Balmanoukian AS, Eder JP, Patnaik A, Aggarwal C, Gubens M, Horn L, Carcereny E, Ahn MJ, Felip E, Lee JS, Hellmann MD, Hamid O, Goldman JW, Soria JC, Dolled-Filhart M, Rutledge RZ, Zhang J, Lunceford JK, Rangwala R, Lubiniecki GM, Roach C, Emancipator K, Gandhi L; KEYNOTE-001 Investigators. Pembrolizumab for the treatment of non-small-cell lung cancer. N Engl J Med. 2015 May 21;372(21):2018-28. doi: 10.1056/NEJMoa1501824. Epub 2015 Apr 19. PMID 25891174
- [Background] Brahmer J, Reckamp KL, Baas P, Crino L, Eberhardt WE, Poddubskaya E, Antonia S, Pluzanski A, Vokes EE, Holgado E, Waterhouse D, Ready N, Gainor J, Aren Frontera O, Havel L, Steins M, Garassino MC, Aerts JG, Domine M, Paz-Ares L, Reck M, Baudelet C, Harbison CT, Lestini B, Spigel DR. Nivolumab versus Docetaxel in Advanced Squamous-Cell Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Jul 9;373(2):123-35. doi: 10.1056/NEJMoa1504627. Epub 2015 May 31. PMID 26028407
- [Background] Borghaei H, Paz-Ares L, Horn L, Spigel DR, Steins M, Ready NE, Chow LQ, Vokes EE, Felip E, Holgado E, Barlesi F, Kohlhaufl M, Arrieta O, Burgio MA, Fayette J, Lena H, Poddubskaya E, Gerber DE, Gettinger SN, Rudin CM, Rizvi N, Crino L, Blumenschein GR Jr, Antonia SJ, Dorange C, Harbison CT, Graf Finckenstein F, Brahmer JR. Nivolumab versus Docetaxel in Advanced Nonsquamous Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Oct 22;373(17):1627-39. doi: 10.1056/NEJMoa1507643. Epub 2015 Sep 27. PMID 26412456
- [Background] Barlesiet al, et al. ESMO 2016 LBA44
- [Background] Reck M, Rodriguez-Abreu D, Robinson AG, Hui R, Csoszi T, Fulop A, Gottfried M, Peled N, Tafreshi A, Cuffe S, O'Brien M, Rao S, Hotta K, Leiby MA, Lubiniecki GM, Shentu Y, Rangwala R, Brahmer JR; KEYNOTE-024 Investigators. Pembrolizumab versus Chemotherapy for PD-L1-Positive Non-Small-Cell Lung Cancer. N Engl J Med. 2016 Nov 10;375(19):1823-1833. doi: 10.1056/NEJMoa1606774. Epub 2016 Oct 8. PMID 27718847
- [Background] Chen N, Fang W, Zhan J, Hong S, Tang Y, Kang S, Zhang Y, He X, Zhou T, Qin T, Huang Y, Yi X, Zhang L. Upregulation of PD-L1 by EGFR Activation Mediates the Immune Escape in EGFR-Driven NSCLC: Implication for Optional Immune Targeted Therapy for NSCLC Patients with EGFR Mutation. J Thorac Oncol. 2015 Jun;10(6):910-23. doi: 10.1097/JTO.0000000000000500. PMID 25658629
- [Background] Jia M, Feng W, Kang S, Zhang Y, Shen J, He J, Jiang L, Wang W, Guo Z, Peng G, Chen G, He J, Liang W. Evaluation of the efficacy and safety of anti-PD-1 and anti-PD-L1 antibody in the treatment of non-small cell lung cancer (NSCLC): a meta-analysis. J Thorac Dis. 2015 Mar;7(3):455-61. doi: 10.3978/j.issn.2072-1439.2015.02.06. PMID 25922725
- [Background] Carbognin L, Pilotto S, Milella M, Vaccaro V, Brunelli M, Calio A, Cuppone F, Sperduti I, Giannarelli D, Chilosi M, Bronte V, Scarpa A, Bria E, Tortora G. Differential Activity of Nivolumab, Pembrolizumab and MPDL3280A according to the Tumor Expression of Programmed Death-Ligand-1 (PD-L1): Sensitivity Analysis of Trials in Melanoma, Lung and Genitourinary Cancers. PLoS One. 2015 Jun 18;10(6):e0130142. doi: 10.1371/journal.pone.0130142. eCollection 2015. PMID 26086854
- [Background] Whilding LM, Maher J. ErbB-targeted CAR T-cell immunotherapy of cancer. Immunotherapy. 2015;7(3):229-41. doi: 10.2217/imt.14.120. PMID 25804476
- [Background] Brentjens RJ, Davila ML, Riviere I, Park J, Wang X, Cowell LG, Bartido S, Stefanski J, Taylor C, Olszewska M, Borquez-Ojeda O, Qu J, Wasielewska T, He Q, Bernal Y, Rijo IV, Hedvat C, Kobos R, Curran K, Steinherz P, Jurcic J, Rosenblat T, Maslak P, Frattini M, Sadelain M. CD19-targeted T cells rapidly induce molecular remissions in adults with chemotherapy-refractory acute lymphoblastic leukemia. Sci Transl Med. 2013 Mar 20;5(177):177ra38. doi: 10.1126/scitranslmed.3005930. PMID 23515080
- [Background] Davila ML, Riviere I, Wang X, Bartido S, Park J, Curran K, Chung SS, Stefanski J, Borquez-Ojeda O, Olszewska M, Qu J, Wasielewska T, He Q, Fink M, Shinglot H, Youssif M, Satter M, Wang Y, Hosey J, Quintanilla H, Halton E, Bernal Y, Bouhassira DC, Arcila ME, Gonen M, Roboz GJ, Maslak P, Douer D, Frattini MG, Giralt S, Sadelain M, Brentjens R. Efficacy and toxicity management of 19-28z CAR T cell therapy in B cell acute lymphoblastic leukemia. Sci Transl Med. 2014 Feb 19;6(224):224ra25. doi: 10.1126/scitranslmed.3008226. PMID 24553386
- [Background] Kochenderfer JN, Dudley ME, Feldman SA, Wilson WH, Spaner DE, Maric I, Stetler-Stevenson M, Phan GQ, Hughes MS, Sherry RM, Yang JC, Kammula US, Devillier L, Carpenter R, Nathan DA, Morgan RA, Laurencot C, Rosenberg SA. B-cell depletion and remissions of malignancy along with cytokine-associated toxicity in a clinical trial of anti-CD19 chimeric-antigen-receptor-transduced T cells. Blood. 2012 Mar 22;119(12):2709-20. doi: 10.1182/blood-2011-10-384388. Epub 2011 Dec 8. PMID 22160384
- [Background] Lee DW, Kochenderfer JN, Stetler-Stevenson M, Cui YK, Delbrook C, Feldman SA, Fry TJ, Orentas R, Sabatino M, Shah NN, Steinberg SM, Stroncek D, Tschernia N, Yuan C, Zhang H, Zhang L, Rosenberg SA, Wayne AS, Mackall CL. T cells expressing CD19 chimeric antigen receptors for acute lymphoblastic leukaemia in children and young adults: a phase 1 dose-escalation trial. Lancet. 2015 Feb 7;385(9967):517-528. doi: 10.1016/S0140-6736(14)61403-3. Epub 2014 Oct 13. PMID 25319501
- [Background] Kochenderfer JN, Dudley ME, Kassim SH, Somerville RP, Carpenter RO, Stetler-Stevenson M, Yang JC, Phan GQ, Hughes MS, Sherry RM, Raffeld M, Feldman S, Lu L, Li YF, Ngo LT, Goy A, Feldman T, Spaner DE, Wang ML, Chen CC, Kranick SM, Nath A, Nathan DA, Morton KE, Toomey MA, Rosenberg SA. Chemotherapy-refractory diffuse large B-cell lymphoma and indolent B-cell malignancies can be effectively treated with autologous T cells expressing an anti-CD19 chimeric antigen receptor. J Clin Oncol. 2015 Feb 20;33(6):540-9. doi: 10.1200/JCO.2014.56.2025. Epub 2014 Aug 25. PMID 25154820
- [Background] Louis CU, Savoldo B, Dotti G, Pule M, Yvon E, Myers GD, Rossig C, Russell HV, Diouf O, Liu E, Liu H, Wu MF, Gee AP, Mei Z, Rooney CM, Heslop HE, Brenner MK. Antitumor activity and long-term fate of chimeric antigen receptor-positive T cells in patients with neuroblastoma. Blood. 2011 Dec 1;118(23):6050-6. doi: 10.1182/blood-2011-05-354449. Epub 2011 Oct 7. PMID 21984804
- [Background] Lamers CH, Sleijfer S, van Steenbergen S, van Elzakker P, van Krimpen B, Groot C, Vulto A, den Bakker M, Oosterwijk E, Debets R, Gratama JW. Treatment of metastatic renal cell carcinoma with CAIX CAR-engineered T cells: clinical evaluation and management of on-target toxicity. Mol Ther. 2013 Apr;21(4):904-12. doi: 10.1038/mt.2013.17. Epub 2013 Feb 19. PMID 23423337
- [Background] Saied A, Licata L, Burga RA, Thorn M, McCormack E, Stainken BF, Assanah EO, Khare PD, Davies R, Espat NJ, Junghans RP, Katz SC. Neutrophil:lymphocyte ratios and serum cytokine changes after hepatic artery chimeric antigen receptor-modified T-cell infusions for liver metastases. Cancer Gene Ther. 2014 Nov;21(11):457-62. doi: 10.1038/cgt.2014.50. Epub 2014 Oct 3. PMID 25277132
- [Background] Gross G, Waks T, Eshhar Z. Expression of immunoglobulin-T-cell receptor chimeric molecules as functional receptors with antibody-type specificity. Proc Natl Acad Sci U S A. 1989 Dec;86(24):10024-8. doi: 10.1073/pnas.86.24.10024. PMID 2513569
- [Background] Eshhar Z, Waks T, Gross G, Schindler DG. Specific activation and targeting of cytotoxic lymphocytes through chimeric single chains consisting of antibody-binding domains and the gamma or zeta subunits of the immunoglobulin and T-cell receptors. Proc Natl Acad Sci U S A. 1993 Jan 15;90(2):720-4. doi: 10.1073/pnas.90.2.720. PMID 8421711
- [Background] Porter DL, Levine BL, Kalos M, Bagg A, June CH. Chimeric antigen receptor-modified T cells in chronic lymphoid leukemia. N Engl J Med. 2011 Aug 25;365(8):725-33. doi: 10.1056/NEJMoa1103849. Epub 2011 Aug 10. PMID 21830940
- [Background] Savoldo B, Ramos CA, Liu E, Mims MP, Keating MJ, Carrum G, Kamble RT, Bollard CM, Gee AP, Mei Z, Liu H, Grilley B, Rooney CM, Heslop HE, Brenner MK, Dotti G. CD28 costimulation improves expansion and persistence of chimeric antigen receptor-modified T cells in lymphoma patients. J Clin Invest. 2011 May;121(5):1822-6. doi: 10.1172/JCI46110. Epub 2011 Apr 11. PMID 21540550
- [Background] Milone MC, Fish JD, Carpenito C, Carroll RG, Binder GK, Teachey D, Samanta M, Lakhal M, Gloss B, Danet-Desnoyers G, Campana D, Riley JL, Grupp SA, June CH. Chimeric receptors containing CD137 signal transduction domains mediate enhanced survival of T cells and increased antileukemic efficacy in vivo. Mol Ther. 2009 Aug;17(8):1453-64. doi: 10.1038/mt.2009.83. Epub 2009 Apr 21. PMID 19384291
- [Background] June CH, Riddell SR, Schumacher TN. Adoptive cellular therapy: a race to the finish line. Sci Transl Med. 2015 Mar 25;7(280):280ps7. doi: 10.1126/scitranslmed.aaa3643. PMID 25810311
- [Background] Morgan RA, Yang JC, Kitano M, Dudley ME, Laurencot CM, Rosenberg SA. Case report of a serious adverse event following the administration of T cells transduced with a chimeric antigen receptor recognizing ERBB2. Mol Ther. 2010 Apr;18(4):843-51. doi: 10.1038/mt.2010.24. Epub 2010 Feb 23. PMID 20179677
- [Background] Dunn GP, Old LJ, Schreiber RD. The immunobiology of cancer immunosurveillance and immunoediting. Immunity. 2004 Aug;21(2):137-48. doi: 10.1016/j.immuni.2004.07.017. PMID 15308095
- [Background] Gajewski TF, Schreiber H, Fu YX. Innate and adaptive immune cells in the tumor microenvironment. Nat Immunol. 2013 Oct;14(10):1014-22. doi: 10.1038/ni.2703. PMID 24048123
- [Background] Zou W, Chen L. Inhibitory B7-family molecules in the tumour microenvironment. Nat Rev Immunol. 2008 Jun;8(6):467-77. doi: 10.1038/nri2326. PMID 18500231
- [Background] Kamphorst AO, Ahmed R. Manipulating the PD-1 pathway to improve immunity. Curr Opin Immunol. 2013 Jun;25(3):381-8. doi: 10.1016/j.coi.2013.03.003. Epub 2013 Apr 9. PMID 23582509
- [Background] Dai S, Jia R, Zhang X, Fang Q, Huang L. The PD-1/PD-Ls pathway and autoimmune diseases. Cell Immunol. 2014 Jul;290(1):72-9. doi: 10.1016/j.cellimm.2014.05.006. Epub 2014 May 27. PMID 24908630
- [Background] Kataoka K, Shiraishi Y, Takeda Y, Sakata S, Matsumoto M, Nagano S, Maeda T, Nagata Y, Kitanaka A, Mizuno S, Tanaka H, Chiba K, Ito S, Watatani Y, Kakiuchi N, Suzuki H, Yoshizato T, Yoshida K, Sanada M, Itonaga H, Imaizumi Y, Totoki Y, Munakata W, Nakamura H, Hama N, Shide K, Kubuki Y, Hidaka T, Kameda T, Masuda K, Minato N, Kashiwase K, Izutsu K, Takaori-Kondo A, Miyazaki Y, Takahashi S, Shibata T, Kawamoto H, Akatsuka Y, Shimoda K, Takeuchi K, Seya T, Miyano S, Ogawa S. Aberrant PD-L1 expression through 3'-UTR disruption in multiple cancers. Nature. 2016 Jun 16;534(7607):402-6. doi: 10.1038/nature18294. Epub 2016 May 23. PMID 27281199
- [Background] Casey SC, Tong L, Li Y, Do R, Walz S, Fitzgerald KN, Gouw AM, Baylot V, Gutgemann I, Eilers M, Felsher DW. MYC regulates the antitumor immune response through CD47 and PD-L1. Science. 2016 Apr 8;352(6282):227-31. doi: 10.1126/science.aac9935. Epub 2016 Mar 10. PMID 26966191
- [Background] Thompson RH, Dong H, Lohse CM, Leibovich BC, Blute ML, Cheville JC, Kwon ED. PD-1 is expressed by tumor-infiltrating immune cells and is associated with poor outcome for patients with renal cell carcinoma. Clin Cancer Res. 2007 Mar 15;13(6):1757-61. doi: 10.1158/1078-0432.CCR-06-2599. PMID 17363529
- [Background] Herbst RS, Soria JC, Kowanetz M, Fine GD, Hamid O, Gordon MS, Sosman JA, McDermott DF, Powderly JD, Gettinger SN, Kohrt HE, Horn L, Lawrence DP, Rost S, Leabman M, Xiao Y, Mokatrin A, Koeppen H, Hegde PS, Mellman I, Chen DS, Hodi FS. Predictive correlates of response to the anti-PD-L1 antibody MPDL3280A in cancer patients. Nature. 2014 Nov 27;515(7528):563-7. doi: 10.1038/nature14011. PMID 25428504
- [Background] Postow MA, Callahan MK, Wolchok JD. Immune Checkpoint Blockade in Cancer Therapy. J Clin Oncol. 2015 Jun 10;33(17):1974-82. doi: 10.1200/JCO.2014.59.4358. Epub 2015 Jan 20. PMID 25605845
- [Background] Riley JL, June CH. The CD28 family: a T-cell rheostat for therapeutic control of T-cell activation. Blood. 2005 Jan 1;105(1):13-21. doi: 10.1182/blood-2004-04-1596. Epub 2004 Sep 7. PMID 15353480
- [Background] Posey AD Jr, Schwab RD, Boesteanu AC, Steentoft C, Mandel U, Engels B, Stone JD, Madsen TD, Schreiber K, Haines KM, Cogdill AP, Chen TJ, Song D, Scholler J, Kranz DM, Feldman MD, Young R, Keith B, Schreiber H, Clausen H, Johnson LA, June CH. Engineered CAR T Cells Targeting the Cancer-Associated Tn-Glycoform of the Membrane Mucin MUC1 Control Adenocarcinoma. Immunity. 2016 Jun 21;44(6):1444-54. doi: 10.1016/j.immuni.2016.05.014. PMID 27332733
- [Background] Chen F, Teachey DT, Pequignot E, Frey N, Porter D, Maude SL, Grupp SA, June CH, Melenhorst JJ, Lacey SF. Measuring IL-6 and sIL-6R in serum from patients treated with tocilizumab and/or siltuximab following CAR T cell therapy. J Immunol Methods. 2016 Jul;434:1-8. doi: 10.1016/j.jim.2016.03.005. Epub 2016 Apr 3. PMID 27049586
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Wolchok JD, Hoos A, O'Day S, Weber JS, Hamid O, Lebbe C, Maio M, Binder M, Bohnsack O, Nichol G, Humphrey R, Hodi FS. Guidelines for the evaluation of immune therapy activity in solid tumors: immune-related response criteria. Clin Cancer Res. 2009 Dec 1;15(23):7412-20. doi: 10.1158/1078-0432.CCR-09-1624. Epub 2009 Nov 24. PMID 19934295
- [Background] Zhao J, Xiong J. [Advances on driver oncogenes of non-small cell lung cancer]. Zhongguo Fei Ai Za Zhi. 2015 Jan;18(1):42-7. doi: 10.3779/j.issn.1009-3419.2015.01.07. Chinese. PMID 25603872

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm: CAR-T cells to treat advanced lung cancer. This study has only one arm. All participators will attend the screening and meet the set criteria for the clinical treatment. PD-L1 CAR-T cells are infused on day 0 with 10%, day 3 with 30% and day 7 with 60% , (1-2)×10^6/kg PD-L1 CAR-T cells total.
  CAR-T cells to treat advanced lung cancer: Drug: fludarabine. On days -4 through -2, fludarabine (25mg/m2) will be infused for 3 consecutive days; Drug: cyclophosphamide. On days -4 through -2, cyclophosphamide (250mg/m2) will be infused for 3 consecutive days.
  Patients will receive the above chemotherapy for lymphocyte-depletion followed by PD-L1 CAR-T cells.
Period: Overall Study
Arm/Group | Treatment Arm
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 1
Age, Customized [Mean (Full Range); unit: years]
  age | 61 [61 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  China | 1
Tumor Stage [Count of Participants; unit: Participants] — Patients tumor staged as IVa with malignant pleural effusion by AJCC Cancer Staging Manual, Eighth Edition (2017).
  Participants | 1
EGFR mutation status [Count of Participants; unit: Participants] — Epidermal growth factor receptor mutation status: wild type
  Participants | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events Associated With PD-L1 CAR-T Cell Treatment
Description: Assessed by the treatment-emergent adverse events as recorded on the case report form, vital signs, laboratory variables, physical examination, electrocardiogram. Treatment-emergent adverse events will be assessed and recorded according to CTCae v4.02.
  No statistical analysis was performed becuase the study was terminated after only 1 patient received treatment.
Time Frame: From the date of CAR-T cell infusion through study completion, average 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 1
Participants | 1

2. Secondary Outcome: Number of Participants Experiencing a Complete (CR) or Partial (PR) Tumor Response
Description: Tumor response will be assessed according to RECIST V1.1. The overall response rate calculated by the numbers of PR or CR / all patients received treatment. The disease control rate calculated by the numbers of CR PR and stable disease / all patients received treatment.
Time Frame: Every three month through study completion, average 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 1
Participants | 1

3. Other Pre Specified Outcome: Numbers of Patients Received Surveillance of PD-L1 CAR-T Cells in Vivo
Description: Using flow cytometry to count of PD-L1 CAR-T cells, calculated the CAR-T cells existence by time after the infusion.
Time Frame: Day 7 after CAR-T cell infusion, and every 2 months up to 2 years
Population: Only 1 patients received treatment and accepted the surveillance of PD-L1 CAR-T cells, and only one detection was performed at Day 7 time point
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 1
Participants | 1

4. Other Pre Specified Outcome: Assessment of Count of the Functional B Cells in Peripheral Blood.
Description: Exploring the correlation of the immune functions of pre- and post-CAR-T cell treatments with the treatment safety and efficacy.
Time Frame: Baseline, day 7 and 30 after the CAR-T cell infusion
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Assessment of Count of the Functional T Cells in Peripheral Blood.
Description: as for outcome 4
Time Frame: Baseline, day 7 and 30 after the CAR-T cell infusion
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 months
Description: Serious Cytokine Release Syndrome causes interstitial pneumonia disease. CTCAE grade 4, possibly drug related.
  Febrile without any courses and respiratory distress that deteriorated quickly into failure in 3 days.He was immediately transferred to the ICU where he received oxygen via nasal cannula and given intravenous infusions of tocilizumab and large doses of methylprednisolone. His symptoms were quickly improved and the pulmonary inflammation became dissipated gradually.
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=1)
interstitial pneumonia disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Serious Cytokine Release Syndrome causes interstitial pneumonia disease. CTCAE grade 4, possibly drug related.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=1)
Serious Cytokine Release Syndrome causes interstitial pneumonia disease. (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Uric acid elevation (Renal and urinary disorders) | 1 (1) — Grade 1, possibly drug not related.
C-Reactive Protein (General disorders) | 1 (1) — Grade 1, possibly drug not related.
proteinuria (Renal and urinary disorders) | 1 (1) — Grade 1, possibly drug not related.
White blood cell counts increasing (Blood and lymphatic system disorders) | 1 (1) — Grade 1, possibly drug not related.
neutrophilic granulocytosis (Blood and lymphatic system disorders) | 1 (1) — Grade 1, possibly drug not related.
upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 1, possibly drug not related.
hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 1, possibly drug not related.
Chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 1, possibly drug not related.
toothache (Skin and subcutaneous tissue disorders) | 1 (1) — Grade 1, possibly drug not related.
anemia (Blood and lymphatic system disorders) | 1 (1) — Grade 1, possibly drug not related.
Albumin decline (General disorders) | 1 (1) — Grade 1, possibly drug not related.
swelling of eye (Eye disorders) | 1 (1) — Grade 1, possibly drug not related.
thrombocytosis (Blood and lymphatic system disorders) | 1 (1) — Grade 1, possibly drug not related.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-12): https://cdn.clinicaltrials.gov/large-docs/34/NCT03330834/Prot_SAP_000.pdf